CLINICAL TRIAL: NCT00012389
Title: A Multicenter, Open-Label, Randomized, Two-Arm Study of Irinotecan (CPT-11) Versus the Combination of Oxaliplatin + Irinotecan (CPT-11) as Second-Line Treatment of Metastatic Colorectal Carcinoma
Brief Title: Irinotecan With or Without Oxaliplatin in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068524; SANOFI-EFC4585
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2002-10

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan; Oxaliplatin

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if irinotecan is more effective with or without oxaliplatin in treating metastatic colorectal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of irinotecan with or without oxaliplatin in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with metastatic colorectal cancer treated with irinotecan with or without oxaliplatin.
* Compare the response rate, time to tumor-related worsening of symptoms, time to disease progression, onset and duration of responses, and duration of disease stabilization in these patients treated with these regimens.
* Compare the safety of these regimens in these patients.

OUTLINE: This is a randomized, open label, multicenter study. Patients are stratified according to Karnofsky performance status (50-60% vs 70-100%), number of metastatic organs involved (1 vs 2 or more), lactic dehydrogenase (no greater than 1.5 times upper limit of normal (ULN) vs greater than 1.5 times ULN), and prior fluorouracil chemotherapy (adjuvant vs first-line treatment for metastatic disease). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive irinotecan IV over 90 minutes on day 1.
* Arm II: Patients receive oxaliplatin IV over 120 minutes followed by irinotecan IV over 30 minutes on day 1.

Courses repeat in each arm every 3 weeks for 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed at 30 days, every 4 weeks for 3 months, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 596 patients (298 per arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum
* Metastatic or recurrent disease that is not amenable to potentially curative treatment
* Progressive or recurrent disease during or after 1, and only 1, regimen of fluorouracil with or without leucovorin calcium or during or within 6 months after adjuvant chemotherapy with fluorouracil and leucovorin calcium

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 50-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT/SGPT no greater than 2 times ULN (no greater than 5 times ULN if liver metastases present)
* Alkaline phosphatase no greater than 2 times ULN (no greater than 5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No unstable angina
* No New York Heart Association class III or IV congestive heart failure
* No serious cardiac arrhythmia
* No history of cardiac toxicity from fluorouracil/leucovorin calcium
* No myocardial infarction within past 6 months

Pulmonary:

* No interstitial pneumonia or extensive and symptomatic fibrosis of the lung

Other:

* No uncontrolled predisposing colonic or small bowel disorder
* No prior chronic enteropathy, chronic diarrhea, or unresolved bowel obstruction/subobstruction
* No diabetes
* No active infection
* No known current peripheral neuropathy
* No concurrent active cancer except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No intolerance of appropriate antiemetics
* No history of anaphylaxis or potential intolerance to atropine sulfate or loperamide
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy
* No prior irinotecan or oxaliplatin
* No other prior chemotherapy agents except fluorouracil with or without leucovorin calcium as first-line therapy for metastatic disease or in the adjuvant setting

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy to non-target lesions allowed
* No prior radiotherapy to target lesions unless disease progression is documented within the radiation port
* At least 3 weeks since prior radiotherapy

Surgery:

* At least 4 weeks since prior major surgical procedure and recovered
* Prior surgery for primary tumor or metastasis allowed

Other:

* At least 30 days since prior investigational drug
* No concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12; Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G. Haller, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (154):
- United States (100):
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - Oncology Center at Providence Park, Mobile, Alabama
  - Arizona Clinical Research Center, Tucson, Arizona
  - Citrus Valley Medical Center, Covina, California
  - California Cancer Care, Inc., Greenbrae, California
  - Tower Hematology Oncology Medical Group, Los Angeles, California
  - Kenmar Research Institute, Los Angeles, California
  - Los Angeles, California
  - Medical Oncology Care Associates, Orange, California
  - P.M.K. Medical Group, Inc., Oxnard, California
  - Cancer and Blood Institute of the Desert, Rancho Mirage, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Colorado Permanente Medical Group, P.C., Denver, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Whittingham Cancer Center, Norwalk, Connecticut
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Comprehensive Cancer Care Specialists of Boca Raton, Boca Raton, Florida
  - Center for Hematology-Oncology, Boca Raton, Florida
  - Southeast Florida Hematology-Oncology Group, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Hematology and Oncology Associates of Jacksonville, Jacksonville, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Lake Heart and Cancer Medical Center, Leesburg, Florida
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - Hematology and Oncology Consultants, P.A., Orlando, Florida
  - Hematology/Oncology Associates, Port Saint Lucie, Florida
  - Oncology & Hematology Associates of West Broward, Tamarac, Florida
  - University Community Hospital, Tampa, Florida
  - Hematology and Oncology Consultants, Titusville, Florida
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Northwest Medical Specialists, P.C., Arlington Heights, Illinois
  - Dreyer Medical Clinic, Aurora, Illinois
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Cancer Care Center, New Albany, Indiana
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Kentuckiana Cancer Institute, Louisville, Kentucky
  - Norton Healthcare Pavilion, Louisville, Kentucky
  - Veterans Affairs Medical Center - Louisville, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - Doctors Hospital of Jefferson, Metairie, Louisiana
  - Stanley Scott Cancer Center, New Orleans, Louisiana
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Medical Center of Boston, Boston, Massachusetts
  - Berkshire Hematology Oncology, P.C., Pittsfield, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Flint, Michigan
  - Parker Hughes Cancer Center, Roseville, Minnesota
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - Missouri Cancer Care, P.C., Saint Charles, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Great Falls Clinic, Great Falls, Montana
  - Western Montana Clinic, Missoula, Montana
  - Somerset Medical Center, Somerville, New Jersey
  - Cooper Cancer Institute, Voorhees Township, New Jersey
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Queens Medical Associates, PC, Fresh Meadows, New York
  - Queens Hospital Center, Jamaica, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Raleigh Hematology/Oncology Associates - Wake Practice, Raleigh, North Carolina
  - Piedmont Hematology-Oncology Associates, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Hematology Oncology Consultants Inc, Columbus, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - Kaiser Permanente - Portland, Portland, Oregon
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - Abington Hematology Oncology Associates, Incorporated, Meadowbrook, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Physicians East - Quadrangle, Greenville, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Erlanger Health Systems, Chattanooga, Tennessee
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - West Clinic, Memphis, Tennessee
  - Memphis Cancer Center, Memphis, Tennessee
  - Tennessee Oncology, P.L.L.C., Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Lone Star Oncology, Austin, Texas
  - Center for Oncology Research and Treatment, Medical City Hospital, Dallas, Texas
  - Baptist Health System Cancer Program, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Hematology-Oncology Associates of Frederiksburg, Inc., Fredericksburg, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Advanced Health Care, Milwaukee, Wisconsin
  - UW Cancer Center Wausau Hospital, Wausau, Wisconsin
  - Irving Cancer Center, Laramie, Wyoming
- Brazil (8):
  - Porto Alegre Hospital, Porto Alegre, Rio Grande do Sul
  - Instituto de Oncologia de Soracaba, Sorocaba, São Paulo
  - Hospital Joao Alves Fiho, Aracaiu-SE
  - Hospital Socor, Belo Horizonte-MG
  - Hospital Erastos Gaertner, Curitiba-PR
  - Instituto Nacional de Cancer, Rio de Janeiro
  - Oncologistas Associados, Rio de Janeiro
  - Hospital do Cancer A C Comargo, São Paulo
- Canada (21):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Royal Victoria Hospital, Barrie, Barrie, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Cite de la Sante de Laval, Laval, Quebec
  - L'Hotel Dieu de Levis, Lévis, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Centre Hospitalier de L'Universitaire de Quebec, Pavillon CHUL, Sainte-Foy, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Zoom International Incoporated, Saint Jerome Quebec
- Czechia (4):
  - Centre of Clinical Oncology and Radiation Oncology, České Budějovice
  - Charles University Hospital, Hradec Králové
  - Onkologicka Klinka A Onkologicka Lab, Prague
  - Fakultni Nemocnice V Motole, Prague
- Hungary (7):
  - Semmelweis University, Budapest
  - National Institute of Oncology, Budapest
  - Fovarosi Onkormanyzat Szent Margit Korhaz, Okologia, Budapest
  - Szent Laszlo Korhaz, Budapest
  - Kozponti Honvedkorhaz I. Belgyogyaszat, Budapest
  - Debreceni Egyetem Onkologiai Tanzek, Debrecen
  - Petz Aladar County Hospital, Gydr
- Poland (4):
  - Maria S. Curie Memorial Institute, Gliwice
  - Jagiellonian University, Krakow (Cracow)
  - Institute of Oncology, Lodz
  - Wielkopolskie Centrum Onkologii Oddzial Chemioterapii, Poznan
- United Kingdom (10):
  - St. Luke's Cancer Center, Guildford, England
  - St. Bartholomew's Hospital, London, England
  - Guy's and St. Thomas' Hospitals NHS Trust, London, England
  - Charing Cross Hospital, London, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Derriford Hospital, Plymouth, England
  - Weston Park Hospital, Sheffield, England
  - Royal Marsden Hospital, Sutton, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland

REFERENCES:
- [Result] Haller DG, Rothenberg ML, Wong AO, Koralewski PM, Miller WH Jr, Bodoky G, Habboubi N, Garay C, Olivatto LO. Oxaliplatin plus irinotecan compared with irinotecan alone as second-line treatment after single-agent fluoropyrimidine therapy for metastatic colorectal carcinoma. J Clin Oncol. 2008 Oct 1;26(28):4544-50. doi: 10.1200/JCO.2008.17.1249. PMID 18824706